CLINICAL TRIAL: NCT03989791
Title: The Clinical Effect of Normal Diet and Absolute Diet on Post-polypectomy Patients: an Open-label, Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NFEC-2017-080
Record Dates: First submitted 2019-06-09; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Polyp Colorectal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absolute diet (Active Comparator)
  Interventions: Dietary Supplement: absolute diet
- Normal diet (Experimental)
  Interventions: Dietary Supplement: normal diet

INTERVENTIONS:
Dietary Supplement: absolute diet — Patients in absolute diet group were fasted from any food with intravenous infusion of 5% glucose and sodium chloride instead in the first 24 hours. Then, the patients will be given soup for the next 24 hours if there was no delayed complication or discomfort during the fasting. Finally, they will gradually transit from soup to normal diet such as porridge, noodles and rice in the third 24 hours.
  Arms: Absolute diet
Dietary Supplement: normal diet — Patients in normal diet group were directly given normal diet such as porridge, noodles and rice as usual after polypectomy. Meanwhile, all the patients in two groups were given PPI for 3 days intravenously and restricted from vigorous exercise for 14 days.
  Arms: Normal diet

SUMMARY:
There is no evidence to prove the impact of post-procedural diet on post-polypectomy bleeding (PPB) or delayed perforation. No relevant study has been conducted and it is yet to be determined if absolute diet is necessary for post-polypectomy patients, and the comparison between normal diet and absolute diet also remains unclear. Therefore, we carried out this randomized controlled study to evaluate and compare tthe clinical effect of different diets on post-polypectomy patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 patient with initial diagnosis of colorectal polyp by colonoscopy;
2. The maximum size of polyp is more than 20mm;
3. The patients underwent single ESD procedure for the polyp and agreed to participate this trial.

Exclusion Criteria:

1. Uncontrollable hypertension or diabetes；
2. Severe comorbidities such as cancer and organ failure etc；
3. Patients who were pregnant;
4. Patients had anticoagulants during perioperative period;
5. Patients with poor compliance. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
postoperative adverse event rate | 14-day after polypectomy
  Postoperative AE includes PPB, post polypectomy electrocoagulation syndrome(PPES) and delayed perforation.

SECONDARY OUTCOMES:
length of stay | 14-day after polypectomy
  calculated by subtracting day of admission from day of discharge.
hospitalization cost | 14-day after polypectomy
  represent the hospital's costs of patients at the hospital